CLINICAL TRIAL: NCT02073994
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation and Expansion, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Orally Administered AG-120 in Subjects With Advanced Solid Tumors, Including Glioma, With an IDH1 Mutation
Brief Title: Study of Orally Administered AG-120 in Subjects With Advanced Solid Tumors, Including Glioma, With an IDH1 Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG120-C-002
Record Dates: First submitted 2014-02-21; First posted 2014-02-28 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cholangiocarcinoma; Chondrosarcoma; Glioma; Other Advanced Solid Tumors
Keywords: chondrosarcoma; cholangiocarcinoma; glioma; advanced solid tumors; IDH1; AG-120
MeSH Terms: conditions — Cholangiocarcinoma; Chondrosarcoma; Glioma | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG-120 (Experimental): AG-120 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Subjects may continue treatment with AG-120 until disease progression, development of other unacceptable toxicity or Investigator discretion.
  Interventions: Drug: AG-120

INTERVENTIONS:
Drug: AG-120 — AG-120 administered continuously as a single agent dosed orally on Days 1 to 28 of a 28-day cycle. Subjects may continue treatment with AG-120 until disease progression or development of other unacceptable toxicity

SUMMARY:
The purpose of this Phase I, multicenter study is to evaluate the safety, pharmacokinetics, pharmacodynamics and clinical activity of AG-120 in advanced solid tumors, including glioma, that harbor an IDH1 mutation. The first portion of the study is a dose escalation phase where cohorts of patients will receive ascending oral doses of AG-120 to determine maximum tolerated dose (MTD) and/or the recommended Phase II dose. The second portion of the study is a dose expansion phase where four arms of patients will receive AG-120 to further evaluate the safety, tolerability, and clinical activity of the recommended Phase II dose. Anticipated time on study treatment is until disease progression, unacceptable toxicity occurs or at Investigator discretion.

ELIGIBILITY:
Key Inclusion Criteria:

1. Dose Escalation

   1. Subjects must have histologically or cytologically confirmed, IDH1 gene-mutated advanced solid tumors, including glioma, that have recurred or progressed following standard therapy, or that have not responded to standard therapy.
   2. Subjects must have evaluable disease by RECIST v1.1 for subjects without glioma or by RANO criteria for subjects with glioma.
2. Dose Expansion: Cholangiocarcinoma

   1. Subjects must have histologically-confirmed diagnosis of IDH1 gene-mutated cholangiocarcinoma Stage II, III, or IV (intra-hepatic, extra-hepatic and perihilar) that is not eligible for curative resection, transplantation, or ablative therapies. Tumors of mixed histology are not allowed.
   2. Cholangiocarcinoma subjects must have progressed following gemcitabine-based regimen.
   3. Cholangiocarcinoma subjects must have radiographically measurable disease in at least one site not previously treated with radiation, chemoembolization, radioembolization, or other local ablative procedures; a new area of tumor progression within or adjacent to a previously-treated lesion, if clearly measurable by a radiologist, is acceptable.
3. Dose Expansion: Chondrosarcoma

   a. Subjects must have IDH1 gene-mutated chondrosarcoma that is either locally advanced or metastatic and not amenable to complete surgical excision.
4. Dose Expansion: Non-enhancing Glioma

   1. Subjects must have progressive glioma that is solely non-enhancing on MRI.
   2. Progression of glioma must have occurred over 12 months or less.
   3. Subject must have available at least 3 prior full sets of scans (not including screening), each separated by at least 2 months with less than or equal to 5 mm slice thickness and up to 1 mm interslice gap on either 2D T2 weighted image, 3D T2 weighted image, or FLAIR.
   4. Subjects must not have had prior surgery (biopsy allowed) or radiation therapy within 6 months of enrollment.
5. Dose Expansion: Solid Tumors Not Otherwise Eligible for the Cholangiocarcinoma, Chondrosarcoma, or Non-enhancing Glioma Cohorts

   1. IDH1 gene-mutated solid tumors refractory to conventional therapy or the subject does not tolerate the conventional therapy
   2. Subjects must have radiographically measurable disease in at least one site not previously treated with radiation, chemoembolization, radioembolization, or other local ablative procedures; a new area of tumor progression within or adjacent to a previously-treated lesion, if clearly measurable by a radiologist, is acceptable.
6. Subject must be ≥18 years of age.
7. Subjects must have documented IDH1 gene-mutated disease based on local test evaluation. (Centralized testing will be performed retrospectively.)
8. Subjects must be amenable to serial peripheral blood sampling, urine sampling, and biopsies during the study.
9. Subject must be able to understand and willing to sign an informed consent. A legally authorized representative may consent on behalf of a subject who is otherwise unable to provide informed consent, if acceptable to and approved by the site and/or site's Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
10. Subjects must have ECOG PS of 0 to 1.
11. Subjects must have expected survival of ≥3 months.
12. Subjects must have adequate bone marrow function as evidenced by:

    1. Absolute neutrophil count ≥1.5 ×109/L;
    2. Hemoglobin >9 g/dL (Subjects are allowed to be transfused to this level)
    3. Platelets ≥ 75 × 109/L.
13. Subjects must have adequate hepatic function as evidenced by:

    1. Serum total bilirubin ≤1.5 × upper limit of normal (ULN), unless considered due to Gilbert's disease or disease involvement following approval by the Medical Monitor;
    2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤2.5 × ULN. For subjects with bone metastases and/or suspected disease-related liver or biliary involvement, ALP must be ≤5 × ULN.
14. Subjects must have adequate renal function as evidenced by:

    a. Serum creatinine ≤2.0 × ULN OR b. Creatinine clearance >40 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR) estimation: (140 - Age) x (weight in kg) x (0.85 if female)/72 x serum creatinine
15. Subjects must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer. (For example, subjects with residual Grade 1 toxicity or stable Grade 2 peripheral neuropathy due to prior chemotherapy are allowed with approval of the Medical Monitor.)
16. Female subjects with reproductive potential must agree to undergo medically supervised pregnancy test prior to starting study drug. The first pregnancy test will be performed at screening (within 7 days prior to first study drug administration), and on the day of the first study drug administration and confirmed negative prior to dosing. Subjects with reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy or tubal occlusion or who have not been naturally postmenopausal (i.e., who have not menstruated at all) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Females of reproductive potential, as well as fertile men with partners who are female of reproductive potential, must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study and for 90 days (females and males) following the last dose of AG-120. A highly effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, double-barrier method (e.g., synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization.

Exclusion Criteria:

1. Subjects who received systemic anticancer therapy or radiotherapy <21 days prior to their first day of study drug administration.
2. Subjects who received an investigational agent <14 days prior to their first day of study drug administration. In addition, the first dose of AG-120 should not occur before a period ≥5 half-lives of the investigational agent has elapsed.
3. Subjects taking the following sensitive cytochrome P450 (CYP) 3A4 substrate medications are excluded from the study unless they can be transferred to other medications prior to enrolling: alfentanil, aprepitant, budesonide, buspirone, conivaptan, darifenacin, darunavir, dronedarone, eletriptan, eplerenone, felodipine, indinavir, fluticasone, lopinavir, lovastatin, lurasidone, maraviroc, midazolam, nisoldipine, quetiapine, saquinavir, sildenafil, simvastatin, tolvaptan, tipranavir, triazolam, ticagrelor, vardenafil and/or the CYP2B6 substrates: bupropion, efavirenz.
4. Subjects taking the following P-glycoprotein (P-gp) transporter-sensitive substrate medications are excluded from the study unless they can be transferred to other medications prior to enrolling: aliskiren, ambrisentan, colchicine, dabigatran etexilate, digoxin, fexofenadine, maraviroc, posaconazole, ranolazine, saxagliptin, sitagliptin, talinolol, and tolvaptan.
5. Subjects for whom potentially curative anticancer therapy is available.
6. Subjects who are pregnant or breast feeding.
7. Subjects with an active severe infection that required anti-infective therapy or with an unexplained fever >38.5°C during screening visits or on their first day of study drug administration (at the discretion of the Investigator, subjects with tumor fever may be enrolled).
8. Subjects with known hypersensitivity to any of the components of AG-120.
9. Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within approximately 28 days of C1D1.
10. Subjects with a history of myocardial infarction within the last 6 months.
11. Subjects with known unstable or uncontrolled angina pectoris.
12. Subjects with a known history of severe and/or uncontrolled ventricular arrhythmias.
13. Subjects with heart-rate corrected QT (QTc) interval ≥ 450 msec or with other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Subjects with right bundle branch block and a prolonged QTc interval should be reviewed by the Medical Monitor for potential inclusion.
14. Subjects taking medications that are known to prolong the QT interval (see Section 9.11.3).
15. Subjects with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C.
16. Subjects with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, or participate in the study.
17. Subjects with known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
18. Subjects with brain metastases that are untreated, symptomatic, or require therapy to control symptoms; or any radiation, surgery, or other therapy, including those used to control symptoms, within 2 months of first dose. Subjects with glioma who are on a stable, steroid dosing regimen 5 days prior to the screening MRI may be permitted to enroll with Medical Monitor approval.
19. Subjects with a history of Grade 4 astrocytoma (applicable only to subjects enrolled in the dose expansion non-enhancing glioma cohort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability: incidence of adverse events | Up to 26 weeks, on average
Maximum Tolerated Dose and/or the recommended Phase II dose of AG-120 in subjects with advanced solid tumors, including glioma | Up to 26 weeks, on average

SECONDARY OUTCOMES:
Dose Limiting Toxicities of AG-120 in subjects with advanced solid tumors, including glioma | Up to 26 weeks, on average
Pharmacokinetics of AG-120 in subjects with advanced solid tumors, including glioma | Up to 26 weeks, on average
  Descriptive statistics will be used to summarize PK parameters for each dose group and, where appropriate, for the entire population. Such parameters will include max concentration (Cmax), time to maximum concentration (Tmax), AUC, elimination half-life.
Pharmacodynamic relationship of AG-120 and 2-HG | Up to 26 weeks, on average
  PD parameters will be summarized using the following descriptive statistics: n, Mean, SD, CV%, Median, Min, and Max, GeoMean, and GeoCV%.
  PK/PD correlations between exposure to AG-120 and the extent of suppression of 2-HG will be explored using graphical display of data.
Clinical Activity associated with AG-120 in subjects with advanced solid tumors, including glioma | Up to 26 weeks, on average
  The clinical activity of AG-120 will be evaluated by assessing response to treatment according to RECIST v1.1 for subjects without glioma or by modified RANO criteria for subjects with glioma

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Scottsdale, Arizona
  - Los Angeles, California
  - Aurora, Colorado
  - Miami, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
- Villejuif, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Tap WD, Cote GM, Burris H, Gore L, Elias A, Beeram M, Conley AP, Gianolio DA, Qu Z, Pandya S, Trent JC. Phase I Study of the Mutant IDH1 Inhibitor Ivosidenib: Long-term Safety and Clinical Activity in Patients with Conventional Chondrosarcoma. Clin Cancer Res. 2025 Jun 3;31(11):2108-2114. doi: 10.1158/1078-0432.CCR-24-4128. PMID 40100120
- [Derived] Ellingson BM, Kim GHJ, Brown M, Lee J, Salamon N, Steelman L, Hassan I, Pandya SS, Chun S, Linetsky M, Yoo B, Wen PY, Mellinghoff IK, Goldin J, Cloughesy TF. Volumetric measurements are preferred in the evaluation of mutant IDH inhibition in non-enhancing diffuse gliomas: Evidence from a phase I trial of ivosidenib. Neuro Oncol. 2022 May 4;24(5):770-778. doi: 10.1093/neuonc/noab256. PMID 34751786
- [Derived] Aguado-Fraile E, Tassinari A, Ishii Y, Sigel C, Lowery MA, Goyal L, Gliser C, Jiang L, Pandya SS, Wu B, Bardeesy N, Choe S, Deshpande V. Molecular and morphological changes induced by ivosidenib correlate with efficacy in mutant-IDH1 cholangiocarcinoma. Future Oncol. 2021 Jun;17(16):2057-2074. doi: 10.2217/fon-2020-1274. Epub 2021 Mar 12. PMID 33709779
- [Derived] Mellinghoff IK, Ellingson BM, Touat M, Maher E, De La Fuente MI, Holdhoff M, Cote GM, Burris H, Janku F, Young RJ, Huang R, Jiang L, Choe S, Fan B, Yen K, Lu M, Bowden C, Steelman L, Pandya SS, Cloughesy TF, Wen PY. Ivosidenib in Isocitrate Dehydrogenase 1-Mutated Advanced Glioma. J Clin Oncol. 2020 Oct 10;38(29):3398-3406. doi: 10.1200/JCO.19.03327. Epub 2020 Jun 12. PMID 32530764
- [Derived] Tap WD, Villalobos VM, Cote GM, Burris H, Janku F, Mir O, Beeram M, Wagner AJ, Jiang L, Wu B, Choe S, Yen K, Gliser C, Fan B, Agresta S, Pandya SS, Trent JC. Phase I Study of the Mutant IDH1 Inhibitor Ivosidenib: Safety and Clinical Activity in Patients With Advanced Chondrosarcoma. J Clin Oncol. 2020 May 20;38(15):1693-1701. doi: 10.1200/JCO.19.02492. Epub 2020 Mar 24. PMID 32208957
- [Derived] Lowery MA, Burris HA 3rd, Janku F, Shroff RT, Cleary JM, Azad NS, Goyal L, Maher EA, Gore L, Hollebecque A, Beeram M, Trent JC, Jiang L, Fan B, Aguado-Fraile E, Choe S, Wu B, Gliser C, Agresta SV, Pandya SS, Zhu AX, Abou-Alfa GK. Safety and activity of ivosidenib in patients with IDH1-mutant advanced cholangiocarcinoma: a phase 1 study. Lancet Gastroenterol Hepatol. 2019 Sep;4(9):711-720. doi: 10.1016/S2468-1253(19)30189-X. Epub 2019 Jul 9. PMID 31300360
- [Derived] Fan B, Mellinghoff IK, Wen PY, Lowery MA, Goyal L, Tap WD, Pandya SS, Manyak E, Jiang L, Liu G, Nimkar T, Gliser C, Prahl Judge M, Agresta S, Yang H, Dai D. Clinical pharmacokinetics and pharmacodynamics of ivosidenib, an oral, targeted inhibitor of mutant IDH1, in patients with advanced solid tumors. Invest New Drugs. 2020 Apr;38(2):433-444. doi: 10.1007/s10637-019-00771-x. Epub 2019 Apr 26. PMID 31028664
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/